CLINICAL TRIAL: NCT05529953
Title: Bioavailability Assays of Oleanolic Acid, Formulated as Functional Olive Oil, in Healthy Subjects. Pharmacokinetic Analysis and Study of Its Integration in Postprandial Human Triglyceride-Rich Lipoproteins
Brief Title: Bioavailability of Oleanolic Acid Formulated as Functional Olive Oil
Acronym: BIO-OLTRAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spanish National Research Council (Other Government)
Collaborators: Andalusian Health Service (Other Government); Universidad Pablo de Olavide (Other)
Responsible Party: Principal Investigator, José M. Castellano, PhD, Principal Investigator, Spanish National Research Council
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PID2019-107837RB-100; PID2019-107837RB-100 (Other Grant/Funding Number: Spanish National Research Agency)
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Healthy Subjects; Bioavailability
Keywords: Oleanolic acid; bioavailability; triglyceride-rich lipoproteins; postprandial dietary intervention; pharmacokinetic; randomized and controlled trial; crossover design
MeSH Terms: interventions — Oleanolic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Double-blind trial. Each recruited participant is assigned a random alphanumeric ID code. Assignment of participants to study groups is done by randomization of their ID.
  The olive oils (functional and control) used in the postprandial trial are labeled with alphanumeric codes known only to the principal investigator of the project.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oleanolic acid-enriched functional olive oil (Experimental): functional olive oil elaborated enriching the control olive oil with Oleanolic acid up to 600 mg OA/kg oil.
  Single oral intake of 55 mL of functional olive oil (dose equivalent to 30 mg OA).
  Interventions: Dietary Supplement: Oleanolic acid (CAS no. 598-02-1; PubChem CID 10494)
- Control olive oil (Active Comparator): commercial olive oil (blend of virgin and refined olive oils) chosen by its very low content of bioactive minor components.
  Single oral intake of 55 mL of commercial olive oil
  Interventions: Dietary Supplement: Control commercial olive oil

INTERVENTIONS:
Dietary Supplement: Oleanolic acid (CAS no. 598-02-1; PubChem CID 10494) — Postprandial study of bioavailability of Oleanolic acid, formulated as functional olive oil, in healthy subjects
  Other Names: Oleanolic acid-enriched functional olive oil
  Arms: Oleanolic acid-enriched functional olive oil
Dietary Supplement: Control commercial olive oil — Postprandial study of Oleanolic acid bioavailability in healthy subjects
  Arms: Control olive oil

SUMMARY:
The oral bioavailability of Oleanolic acid (OA) when formulated as functional olive oil, and its mechanisms of systemic transport, will be approached by mean of randomized and controlled trial with 20 healthy volunteers. Ten individuals randomly selected will receive 55 mL of the functional OA-enriched olive oil (equivalent dose 30 mg OA) as part of an experimental breakfast. The other ten participants will receive within this experimental meal the same amount of the control olive oil. Immediately before and after eating the respective breakfasts, aliquots of cubital blood will be drawn every hour, over a postprandial period of 7 hours. Since in this trial design, each participant is his/her own control, a four-week washout period is established, after which a new series of tests that cross the type of olive oil consumed will be carried out.

From the aliquots of cubital blood, sera will be obtained by centrifugation. The extraction and quantification of serum OA will be realized by gas chromatography (GC) using flame ionization (FID) and mass spectrometry (MS) detectors. In the pharmacokinetic analysis of data, a mono-compartmental model will be assumed. It will be determined: 1) absorption parameters such as the maximum concentration achieved and the timing for it, the constant of absorption and the area under the curve; 2) distribution parameters such as the constant and volume of distribution; 3) metabolism parameters, such as the OA fraction associated with albumin; and 4) elimination parameters such as the elimination constant, the half-life and the clearance.

To demonstrate the presence of OA in postprandial TRL, chylomicron and VLDL fractions will be prepared by plasma ultrafiltration in normal saline, and hydrolysed with pancreatic enzyme. The possible presence of OA among the TRL-derived lipids will be evaluated. The content of apo B48 and B100, as markers of the presence of chylomicrons and VLDL, respectively, will be determined by ELISA.

Other parameters related to glycemic control, such as serum insulin, C-peptide and GLP-1 will be analyzed by ELISA.

DETAILED DESCRIPTION:
Design and implementation of the biovailability assays The study of oral bioavailability of Oleanolic acid (OA) when formulated as functional olive oil, and its mechanisms of systemic transport, will be approached by mean of a postprandial intervention with 20 healthy volunteers.

The participants will be recruited after the complete biochemical and hematological analysis yield results within normal limits, and after checking in their electronic medical histories that they do not suffer from digestive, metabolic or oncologic disorders or any other pathology that, in opinion of the clinical investigators, could prevent them from participating in the trial. For their inclusion in the trial, it is also required that they grant the written consent to the protocols approved by the Institutional Committees for Human Research, after being conveniently informed both orally and documentally.

The fieldwork will be performed in the Day Hospital of the Endocrinology and Nutrition Service of the University Hospitals 'Virgen del Rocio' from Seville (SPAIN).

Sample size. The main quantitative variable to be examined in this trial is OA serum concentration. In the absence of consistent baseline data published so far, data from the analysis of OA in sera of the PREDIABOLE Study (ISRCTN03372660) have been used. A cohort of 25 participants from the control group, consuming commercial olive oil, was selected, and an average baseline concentration of 155 ± 72 ng OA/mL was determined. Considering this, it is now postulated that the plasma OA content will increase by at least 50% as consequence of the intake of the functional olive oil (equivalent dose 30 mg OA). To prove this unilateral hypothesis test, with a confidence level of 90% (risk α=0.01, zα=1.645) and a power of 95% (zβ=1.645), a sample size of at least 17 volunteers is required. Assuming that losses lower than 15% are tolerable, the adjusted sample size would be 20 subjects.

Anamnesis and physical examination of participants. The anamnesis will include vital data and general history collecting all the symptoms that the individual may present, their medical and surgical history, as well as pharmacological treatments followed. Information about lifestyle, perception of the own body image, diet and kind and intensity of physical activity will be also obtained. In addition, the muscle mass, fatty compartment (adipose panniculus), existence of edema, etc. will be examined. Likewise, systolic and diastolic blood pressure and heart rate will be determined.

Anthropometric study and body composition. The anthropometric study will include the determination of total body weight, height, body mass index (BMI), as well as waist and hip circumferences. The study and evaluation of these variables will be carried out in accordance with the guidelines of the International Society for the Advancement of kinanthropometry (ISAK). The study of body composition will be carried out by electrical bioimpedance, using a TANITA® body composition analyzer model BC-418MA. Fat mass, lean mass, muscle mass, total water, bone mass, basal metabolism and visceral fat will be quantified with this technique, making use of prediction equations validated and adjusted by age and sex.

Biochemical studies. Samples of fasting cubital blood will be drawn to determine the parameters of general, hepatic and renal biochemistry. In addition, a complete urine analysis will be performed, which include the habitual physical, chemical and microscopically measurements. These determinations will be carried out at the Laboratory of Analysis and Clinical Biochemistry of 'Virgen del Rocío' University Hospitals of Seville.

Intervention The participants will be encouraged to avoid the consumption of alcoholic beverages and tobacco during the day preceding the execution of the assays. On trial days, and after 12 hours of overnight fasting, blood samples will be drawn from the cubital vein. Subsequently, ten individuals randomly selected will receive 55 mL of the functional OA-enriched olive oil (equivalent dose 30 mg OA) as part of an experimental breakfast, that includes coffee, skimmed milk and whole-grain toast. The other ten participants will receive within the experimental meal the same amount of the control olive oil. After eating the respective breakfasts, aliquots of cubital blood will be drawn every hour, over a postprandial period of 7 hours. During this time, free access to water intake will be allowed.

A four-week washout period is established, after which a new series of tests that cross the type of olive oil consumed will be carried out.

Pharmacokinetic study of OA From the aliquots of cubital blood, sera will be obtained by centrifugation, and NaN3, PMSF and aprotinin will be added as preservatives, to avoid their proteolytic degradation. Serum samples will be stored at -80 0C in the laboratories of the IG-CSIC until analysis. The extraction and fractionation of serum OA will be realized by liquid/liquid and solid phase extractions, whereas the identification and quantification of the triterpene will be completed by GC-FID and GC-MS. In the pharmacokinetic analysis of data, a mono-compartmental model will be assumed. From data of the serum contents of free OA throughout the postprandial period the following parameters will be determined: 1) absorption parameters such as the maximum concentration achieved and the timing for it, the constant of absorption and the area under the curve; 2) distribution parameters such as the constant and volume of distribution; 3) metabolism parameters, such as the OA fraction associated with albumin; and 4) elimination parameters such as the elimination constant, the half-life and the clearance. For calculations, the SigmaPLot pharmacokinetic analysis module (Systat Software Inc., San Jose, CA, USA) will be used.

Study of the presence of OA in triglyceride rich lipoproteins (TRL). Chylomicrons will be first isolated from plasma in normal saline by centrifugation at 100,000 × g for 20 min. Very low density lipoproteins (VLDL) will be subsequently separated at 230,000 × g for 18 h. The chylomicron and VLDL fractions will be hydrolyzed with pancreatic enzyme. The released lipids will be extracted with chloroform:methanol (2:1), and fractionated by solid/liquid extraction with methanol:chloroform (1:1) and isopropanol:acetonitrile:water (2:1:1). The free fatty acids (FFA) composition will be analysed by GC-FID as the correspondent methyl esters. The possible presence of OA among the TRL-derived lipids will be evaluated after fractionation and GC-MS analysis. The content of apo B48 and B100, as markers of the presence of chylomicrons and VLDL, respectively, will be determined by ELISA.

Other biochemical parameters serum insulin, C-peptide and GLP-1 will be analyzed by ELISA.

ELIGIBILITY:
Inclusion Criteria:

* healthy women and men
* aged 18-30 years
* BMI in the range 18.5-29.9 kg/m2
* complete biochemical and hematological analysis yield results within normal limits
* grant the written consent to the protocols approved by the Institutional Committees for Human Research of the CSIC and HUVR, after being conveniently informed both orally and documentally.

Exclusion Criteria:

* suffering from digestive, metabolic or oncologic disorders or any other pathology that, in opinion of the clinical investigators, could prevent them from participating in the trial (checked in their electronic medical histories).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration Versus Time Curve (AUC) of Oleanolic acid | postpradial 6-hours period
  Quantification of the Oleanolic acid plasma concentration every 60 minutes
Identification and quantification of the Oleanolic acid presence in triglyceride-rich lipoproteins | postpradial 6-hours period
  isolation and analysis of Oleanolic acid in postprandial chylomicrons and VLDL

SECONDARY OUTCOMES:
Fraction of the Oleanolic acid associated to serum albumin | postpradial 6-hours period
  Spectrophotometric analysis of the Oleanolic acid-serum albumin complexes
Influence of the Oleanolic acid-based intervention on the postprandial glycemic control | postpradial 6-hours period
  Determination of glycaemia, insulin, C-peptide and GLP-1
Influence of the Oleanolic acid-based intervention on plasma lipids | postpradial 6-hours period
  Determination of circulating triglycerides, total cholesterol, LDL, HDL

CONTACTS AND LOCATIONS:
Overall Officials: José M. Castellano, PhD, Principal Investigator — Instituto de la Grasa-Spanish National Research Council (CSIC); Pedro P. García-Luna, Principal Investigator — Andalusian Public Foundation for Health Research Management in Seville
Locations (1):
- Universitary Hospitals Virgen del Rocío, Seville, Sevilla, Spain

IPD SHARING:
Plan to Share IPD: No
The datasets generated during the trial are available from the Principal Investigator upon reasonable request.

REFERENCES:
- [Background] Guinda A, Rada M, Delgado T, Gutierrez-Adanez P, Castellano JM. Pentacyclic triterpenoids from olive fruit and leaf. J Agric Food Chem. 2010 Sep 8;58(17):9685-91. doi: 10.1021/jf102039t. PMID 20712364
- [Background] Castellano JM, Guinda A, Delgado T, Rada M, Cayuela JA. Biochemical basis of the antidiabetic activity of oleanolic acid and related pentacyclic triterpenes. Diabetes. 2013 Jun;62(6):1791-9. doi: 10.2337/db12-1215. PMID 23704520
- [Background] Castellano JM, Ramos-Romero S, Perona JS. Oleanolic Acid: Extraction, Characterization and Biological Activity. Nutrients. 2022 Jan 31;14(3):623. doi: 10.3390/nu14030623. PMID 35276982
- [Background] Fernandez-Aparicio A, Correa-Rodriguez M, Castellano JM, Schmidt-RioValle J, Perona JS, Gonzalez-Jimenez E. Potential Molecular Targets of Oleanolic Acid in Insulin Resistance and Underlying Oxidative Stress: A Systematic Review. Antioxidants (Basel). 2022 Aug 3;11(8):1517. doi: 10.3390/antiox11081517. PMID 36009236
- [Background] Santos-Lozano JM, Rada M, Lapetra J, Guinda A, Jimenez-Rodriguez MC, Cayuela JA, Angel-Lugo A, Vilches-Arenas A, Gomez-Martin AM, Ortega-Calvo M, Castellano JM. Prevention of type 2 diabetes in prediabetic patients by using functional olive oil enriched in oleanolic acid: The PREDIABOLE study, a randomized controlled trial. Diabetes Obes Metab. 2019 Nov;21(11):2526-2534. doi: 10.1111/dom.13838. Epub 2019 Aug 28. PMID 31364228
- [Background] Jimenez-Sanchez A, Martinez-Ortega AJ, Remon-Ruiz PJ, Pinar-Gutierrez A, Pereira-Cunill JL, Garcia-Luna PP. Therapeutic Properties and Use of Extra Virgin Olive Oil in Clinical Nutrition: A Narrative Review and Literature Update. Nutrients. 2022 Mar 31;14(7):1440. doi: 10.3390/nu14071440. PMID 35406067
- [Background] Rada M, Castellano JM, Perona JS, Guinda A. GC-FID determination and pharmacokinetic studies of oleanolic acid in human serum. Biomed Chromatogr. 2015 Nov;29(11):1687-92. doi: 10.1002/bmc.3480. Epub 2015 May 5. PMID 25943913
- [Background] Karpe F, Tornvall P, Olivecrona T, Steiner G, Carlson LA, Hamsten A. Composition of human low density lipoprotein: effects of postprandial triglyceride-rich lipoproteins, lipoprotein lipase, hepatic lipase and cholesteryl ester transfer protein. Atherosclerosis. 1993 Jan 4;98(1):33-49. doi: 10.1016/0021-9150(93)90221-f. PMID 8457249